CLINICAL TRIAL: NCT00479466
Title: A Multicenter, Double-Blind, Randomized, Placebo and Active Comparator Controlled Dose-Range Finding Study of MK0893 in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: Dose-Range Finding Study for MK0893 (0893-008)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sufficient data regarding the dose-response to MK-0893 had been obtained from the first cohort of the study to assess the safety and efficacy
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0893-008; 2007_526
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Results first posted 2011-11-11 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — N-((4-(1-(3-(3,5-dichlorophenyl)-5-(6-methoxynaphthalen-2-yl)-1H-pyrazol-1-yl)ethyl)phenyl)carbonyl)-beta-alanine; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- MK0893 80 mg (Experimental): MK0893 tablets totaling 80 mg once daily.
  Interventions: Drug: MK0893; Drug: Placebo to MK0893; Drug: Placebo to Metformin
- MK0893 60 mg (Experimental): MK0893 tablets totaling 60 mg once daily.
  Interventions: Drug: MK0893; Drug: Placebo to MK0893; Drug: Placebo to Metformin
- MK0893 40 mg (Experimental): MK0893 40 mg tablet once daily.
  Interventions: Drug: MK0893; Drug: Placebo to MK0893; Drug: Placebo to Metformin
- MK0893 20 mg (Experimental): MK0893 20 mg tablet once daily.
  Interventions: Drug: MK0893; Drug: Placebo to MK0893; Drug: Placebo to Metformin
- Metformin (Active Comparator): Metformin HCL 500 mg tablet twice daily BID titrating up to 1000 mg twice daily over 3 weeks.
  Interventions: Drug: Metformin; Drug: Placebo to MK0893
- Placebo (Placebo Comparator): PLA tablets. 12 week treatment period.
  Interventions: Drug: Placebo to MK0893; Drug: Placebo to Metformin

INTERVENTIONS:
Drug: MK0893 — MK0893 taken orally once daily; 20 mg and 40 mg tablets used in combination according to dose.
  Arms: MK0893 20 mg; MK0893 40 mg; MK0893 60 mg; MK0893 80 mg
Drug: Metformin — Metformin HCL 500 mg tablet twice daily titrating up to 1000 mg twice daily over 3 weeks.
  Arms: Metformin
Drug: Placebo to MK0893 — Dose-matched placebo tablets to MK0893; taken orally once daily.
Drug: Placebo to Metformin — Dose-matched placebo tablets to metformin (500 mg); taken orally twice daily.
  Arms: MK0893 20 mg; MK0893 40 mg; MK0893 60 mg; MK0893 80 mg; Placebo

SUMMARY:
A study to compare MK0893 to metformin or placebo for patients with Type 2 diabetes (Diabetes Mellitus).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have Type 2 Diabetes Mellitus, with suboptimal glucose control, while either not on AHA (antihyperglycemic agent) therapy or on monotherapy or on low-dose combination therapy

Exclusion Criteria:

* Patients have a history of Type 1 Diabetes Mellitus
* Patients taking insulin or thiazolidinedione (TZD, a peroxisome proliferator-activated receptor [PPAR]-gamma agonist)
* Patients who have a contraindication to metformin

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | MK0893 20 mg | MK0893 40 mg | MK0893 60 mg | MK0893 80 mg | Metformin HCL
Started | 57 | 57 | 57 | 58 | 56 | 57
Completed | 44 | 49 | 54 | 55 | 48 | 53
Not Completed | 13 | 8 | 3 | 3 | 8 | 4
Not completed — Adverse Event | 5 | 1 | 0 | 1 | 2 | 0
Not completed — Hyperglycemia | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 2 | 2
Not completed — Physician Decision | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 5 | 0 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MK0893 20 mg | MK0893 40 mg | MK0893 60 mg | MK0893 80 mg | Metformin HCL | Total
Number analyzed (Participants) | 57 | 57 | 57 | 58 | 56 | 57 | 342
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (10.2) | 55.6 (8.2) | 53.7 (8.2) | 56.1 (7.9) | 53.5 (10.4) | 55.1 (8.2) | 54.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 22 | 26 | 31 | 30 | 168
  Male | 26 | 29 | 35 | 32 | 25 | 27 | 174

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Fasting Plasma Glucose (FPG)
Time Frame: Week 12
Population: All participants who received at least one dose of study therapy, had a baseline measurement, and had at least one post-randomization measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | MK0893 20 mg | MK0893 40 mg | MK0893 60 mg | MK0893 80 mg | Metformin HCL
Number analyzed (Participants) | 54 | 55 | 57 | 57 | 54 | 57
mg/dL | -1.8 [-11.4 to 7.8] | -32.4 [-41.7 to -23.2] | -48.4 [-57.4 to -39.5] | -53.0 [-61.9 to -44.1] | -63.0 [-72.4 to -53.7] | -37.3 [-46.3 to -28.4]
Statistical Analysis 1: Comparison: Placebo vs MK0893 20 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -30.6, 95% CI 2-sided [-44.0 to -17.3]
Statistical Analysis 2: Comparison: Placebo vs MK0893 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -46.6, 95% CI 2-sided [-59.7 to -33.4]
Statistical Analysis 3: Comparison: Placebo vs MK0893 60 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -51.1, 95% CI 2-sided [-64.3 to -38.0]
Statistical Analysis 4: Comparison: Placebo vs MK0893 80 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -61.2, 95% CI 2-sided [-74.6 to -47.8]
Statistical Analysis 5: Comparison: Placebo vs Metformin HCL; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -35.5, 95% CI 2-sided [-48.6 to -22.4]

2. Secondary Outcome: Change From Baseline to Week 12 in Hemoglobin A1c (HbA1c)
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | MK0893 20 mg | MK0893 40 mg | MK0893 60 mg | MK0893 80 mg | Metformin HCL
Number analyzed (Participants) | 48 | 51 | 57 | 57 | 52 | 56
mg/dL | 0.54 [0.27 to 0.82] | -0.60 [-0.87 to -0.33] | -0.99 [-1.25 to -0.73] | -1.14 [-1.40 to -0.89] | -1.52 [-1.79 to -1.25] | -0.78 [-1.04 to -0.52]
Statistical Analysis 1: Comparison: Placebo vs MK0893 20 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-1.53 to -0.76]
Statistical Analysis 2: Comparison: Placebo vs MK0893 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.53, 95% CI 2-sided [-1.91 to -1.15]
Statistical Analysis 3: Comparison: Placebo vs MK0893 60 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.69, 95% CI 2-sided [-2.07 to -1.31]
Statistical Analysis 4: Comparison: Placebo vs MK0893 80 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -2.06, 95% CI 2-sided [-2.45 to -1.68]
Statistical Analysis 5: Comparison: Placebo vs Metformin HCL; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.32, 95% CI 2-sided [-1.70 to -0.95]

3. Secondary Outcome: Change From Baseline to Week 12 in 2-Hour Post Prandial Glucose (PPG)
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | MK0893 20 mg | MK0893 40 mg | MK0893 60 mg | MK0893 80 mg | Metformin HCL
Number analyzed (Participants) | 41 | 47 | 55 | 54 | 47 | 53
mg/dL | -8.1 [-24.6 to 8.4] | -64.9 [-80.3 to -49.5] | -78.1 [-92.4 to -63.8] | -95.5 [-110.0 to -80.9] | -109.7 [-125.1 to -94.3] | -68.9 [-83.4 to -54.3]
Statistical Analysis 1: Comparison: Placebo vs MK0893 20 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -56.8, 95% CI 2-sided [-79.4 to -34.3]
Statistical Analysis 2: Comparison: Placebo vs MK0893 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -70.0, 95% CI 2-sided [-91.8 to -48.2]
Statistical Analysis 3: Comparison: Placebo vs MK0893 60 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -87.4, 95% CI 2-sided [-109.4 to -65.3]
Statistical Analysis 4: Comparison: Placebo vs MK0893 80 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -101.6, 95% CI 2-sided [-124.2 to -79.1]
Statistical Analysis 5: Comparison: Placebo vs Metformin HCL; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -60.8, 95% CI 2-sided [-82.7 to -38.8]

ADVERSE EVENTS:
Arm/Group | Placebo | MK0893 20 mg | MK0893 40 mg | MK0893 60 mg | MK0893 80 mg | Metformin HCL
Serious Adverse Events (participants affected / at risk) | 5/57 | 0/57 | 1/57 | 0/58 | 2/56 | 0/57
Other Adverse Events (participants affected / at risk) | 16/57 | 11/57 | 22/57 | 16/58 | 12/56 | 13/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | MK0893 20 mg (N=57) | MK0893 40 mg (N=57) | MK0893 60 mg (N=58) | MK0893 80 mg (N=56) | Metformin HCL (N=57)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | MK0893 20 mg (N=57) | MK0893 40 mg (N=57) | MK0893 60 mg (N=58) | MK0893 80 mg (N=56) | Metformin HCL (N=57)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 4 (9)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (3) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 5 (6) | 1 (1) | 4 (5) | 5 (7) | 1 (1) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Sufficient data regarding the dose-response to MK-0893 had been obtained from the first cohort of the study to assess the safety and efficacy, thus the study was discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less